CLINICAL TRIAL: NCT03624192
Title: A Prospective Multicenter Randomized Controlled Clinical Study to Investigate the Safety and Effectiveness of RES (Regenerative Epidermal Suspension) Prepared With the RECELL® Device Compared to Conventional Care for Healing of Donor Sites in Infants, Children and Adolescents (Aged 1-16 Years)
Brief Title: RES Prepared With RECELL® Compared to Conventional Care for Healing of Donor Sites in Ages 1-16 Years
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed in response to COVID-19 and overall program objectives.
Sponsor: Avita Medical (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTP006-1
Record Dates: First submitted 2018-07-20; First posted 2018-08-10 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Skin; Deformity
Keywords: Pediatric, Complex Skin Deformities
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Intervention Model Description: Each subject serves as their own control.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RECELL® Autologous Cell Harvesting Device (Experimental): RECELL + Telfa™ Clear and Xeroform™ dressings
  Interventions: Device: RECELL® Autologous Cell Harvesting Device
- Telfa™ Clear and Xeroform™ dressings (Active Comparator): Telfa™ Clear and Xeroform™ dressings
  Interventions: Other: Telfa™ Clear and Xeroform™ dressings

INTERVENTIONS:
Device: RECELL® Autologous Cell Harvesting Device — Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Other Names: RES (Regenerative Epidermal Suspension)
  Arms: RECELL® Autologous Cell Harvesting Device
Other: Telfa™ Clear and Xeroform™ dressings — Telfa™ Clear and Xeroform™ dressings
  Other Names: Control
  Arms: Telfa™ Clear and Xeroform™ dressings

SUMMARY:
To evaluate whether the time to complete closure is superior for RECELL-treated split-thickness donor sites, compared with Control (standardized dressings only). The mean time for donor site healing will be compared between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 1 through 16 years (inclusive) with a skin defect for which autografting is indicated.
2. The area of total injury or planned defect (excluding donor sites) is 5% to 25% Total Body Surface Area (TBSA), inclusive.
3. Two discrete donor sites of similar size (± 25%) can be created in a similar non-articulating location (excluding the scalp) with each donor site representing a minimum of 1% TBSA.
4. The patient and family member/parent/guardian are able to complete all follow-up evaluations required by the study protocol.
5. In the opinion of the Investigator, the patient and/or parent/guardian must be able to:

   1. Understand the full nature and purpose of the study, including possible risks and adverse events, and
   2. Provide informed consent/assent as appropriate for study participation.
6. The patient and/or parent/guardian agrees to abstain from any other treatment of the wound(s) for the duration of the study unless medically necessary and comply with all compulsory study procedures.
7. The patient and/or parent/guardian agrees to abstain from enrollment in any other interventional clinical trial for the duration of the study.
8. The patient and/or parent/guardian can read and understand instructions and give informed, voluntary, written consent.
9. Life expectancy greater than 52 weeks.

Exclusion Criteria:

1. Prior autograft harvest at planned study donor sites.
2. Patients with sepsis or hemodynamic instability.
3. The patient has an infection under active management or other dermatologic condition at the planned donor sites or treatment areas.
4. Patient (of reasonable age) or parent/guardian is unable to follow the protocol requirements.
5. The patient has other concurrent conditions that in the opinion of the Investigator may compromise patient safety or study objectives.
6. Patients with a known hypersensitivity to trypsin or compound sodium lactate for irrigation.
7. In post-pubescent girls, pregnant or breast-feeding (pregnancy test should be performed in accordance with local institutional requirements).
8. Enrollment in a concurrent study in which the study treatment may confound the endpoints of this study.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arizona Burn Center at Maricopa Intergrated Health Systems, Phoenix, Arizona
  - Shriners Hospital for Children, Northern California, Sacramento, California
  - University of California at San Diego, San Diego, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Shriners Hospital for Children, Boston, Boston, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - University of Washington Regional Burn Center at Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Every subject received both interventions (RECELL and CONTROL) such that each subject served as their own control.
  RECELL + Telfa™ Clear and Xeroform™ dressings
  RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Telfa™ Clear and Xeroform™ dressings: Telfa™ Clear and Xeroform™ dressings
Units Other Than Participants: Donor site
Groups:
- RECELL: Every subject received both interventions (RECELL and CONTROL) such that each subject served as their own control.
  RECELL + Telfa™ Clear and Xeroform™ dressings
  RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Telfa™ Clear and Xeroform™ dressings: Telfa™ Clear and Xeroform™ dressings
- Control: very subject received both interventions (RECELL and CONTROL) such that each subject served as their own control.
  RECELL + Telfa™ Clear and Xeroform™ dressings
  RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Telfa™ Clear and Xeroform™ dressings: Telfa™ Clear and Xeroform™ dressings
Period: Overall Study
Arm/Group | RECELL | Control
Started | 3; 3 Donor site | 3; 3 Donor site
Completed | 2; 2 Donor site | 2; 2 Donor site
Not Completed | 1; 1 Donor site | 1; 1 Donor site
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: All Participants (Within Patient Control): All subjects receive both RECELL and Control. Each subject serves as their own control.
Arm/Group | Experimental: All Participants (Within Patient Control)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.7 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Closure
Description: The primary effectiveness endpoint is time, in days, to complete closure (≥95% epithelialization by blinded assessor) of study donor sites confirmed at two consecutive visits.
Time Frame: up to 4 weeks
Measure: Number; unit: Days
Units Other Than Participants: Site
Groups:
- Control: Every subject received both interventions (RECELL and CONTROL) such that each subject served as their own control.
  RECELL + Telfa™ Clear and Xeroform™ dressings
  RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Telfa™ Clear and Xeroform™ dressings: Telfa™ Clear and Xeroform™ dressings
Arm/Group | RECELL | Control
Number analyzed (Participants) | 3 | 3
Number analyzed (Site) | 3 | 3
Days
  Subject 001 | 10 | 10
  Subject 003 | 14 | 11
  Subject 004 | 13 | 13

2. Secondary Outcome: Donor Site Treatment Preference (Site A or Site B) Reported by Subject
Description: Subject will be asked which donor site (A or B) they prefer (if subject is less than 8 years of age parents will be asked)
Time Frame: 4 weeks
Measure: Number; unit: Participants
Groups:
- All Participants: Treatment: RECELL + Telfa™ Clear and Xeroform™ dressings. RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Control: Telfa and Xeroform only
Arm/Group | All Participants
Number analyzed (Participants) | 3
Participants
  RECELL | 1
  Control | 1
  No Response | 1

3. Secondary Outcome: Donor Site Treatment Preference (Site A or Site B) Reported by Physician
Description: Physician will be asked which donor site (A or B) they prefer
Time Frame: 4 weeks
Measure: Number; unit: Physician Response
Arm/Group | All Participants
Number analyzed (Participants) | 3
Physician Response
  RECELL | 1
  Control | 0
  Unable to determine/no preference | 2

4. Secondary Outcome: Comparative Itching of Study Donor Sites Performed by Asking the Child Which Donor Site (A or B) Was Itchier After Treatment
Description: Comparative Itching of study donor sites during 1st week post treatment by asking which site was itchier after treatment
Time Frame: Day 7
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 3
Participants
  RECELL | 0
  Control | 0
  No difference/Can't tell | 3

5. Secondary Outcome: Comparative Pain of Study Donor Sites Performed by Asking the Child Which Donor Site (A or B) Was More Painful Since Treatment
Description: Comparative pain of study donor sites during 1st week post treatment by asking the child which site was more painful since treatment
Time Frame: Day 7 or 8
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 3
Participants
  RECELL | 0
  Control | 0
  No Pain at Either Donor SIte | 1
  No Difference/Can't Tell | 2

6. Secondary Outcome: Blinded Evaluator Overall Opinion Score (1-10) Using the Patient and Observer Scar Assessment Scale (POSAS)
Description: Blinded Evaluator Overall Opinion POSAS Score of study donor sites. The Overall Opinion Score uses a 10-point scale where 10 corresponds to the worst imaginable scar.
Time Frame: Week 24
Population: Data was not collected for subject 001
Measure: Number; unit: Score on a scale
Arm/Group | RECELL | Control
Number analyzed (Participants) | 2 | 2
Score on a scale
  Subject 001: number analyzed (Participants) | 0 | 0
  Subject 003: number analyzed (Participants) | 1 | 1
  Subject 003 | 2 | 9
  Subject 004: number analyzed (Participants) | 1 | 1
  Subject 004 | 2 | 3

7. Secondary Outcome: Patient Overall Opinion Score (1-10) Using the Patient and Observer Scar Assessment Scale (POSAS)
Description: Patient Overall Opinion POSAS Score of study donor sites(reported by subject 8 years of age or older, or by parent/guardian if subject less than 8 years of age). The Overall Opinion Score uses a 10-point scale where 10 corresponds to the worst imaginable scar.
Time Frame: Week 24
Population: Data was not collected from subjects 001 and 004
Measure: Number; unit: Score on a scale
Arm/Group | RECELL® Autologous Cell Harvesting Device | Telfa™ Clear and Xeroform™ Dressings
Number analyzed (Participants) | 1 | 1
Score on a scale
  Subject 001: number analyzed (Participants) | 0 | 0
  Subject 003 | 5 | 10
  Subject 004: number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Investigator's (Unblinded) Assessment of Healing at All RECELL-treated Areas by Direct Observation
Description: Investigator's (unblinded) assessment of healing at all RECELL-treated areas including study donor sites by direct observation
Time Frame: Through Week 52
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mean Subject Reported Pain Score Before and After Dressing Changes
Description: Mean subject (or parent/guardian) reported study donor site pain prior to and after dressing changes. Faces Pain Scale-Revised (FPS-R) or Numeric Rated Pain Scale will be used based on the child's age. Both scales use a 10-point scale where 10 is the worst pain imaginable or very much pain.
Time Frame: Up to Week 4
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Subject Reported Study Donor Site Itching Score Prior to Dressing Changes
Description: Mean subject (or parent/guardian) reported study donor site itching score prior to dressing changes using the Itch Man Scale (0-4) where 4 represents itching most terribly
Time Frame: Up to Week 4
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Health Care Provider's Mean Pain Score Associated With Dressing Changes at Study Donor Sites
Description: Mean pain score associated with dressing changes at study donor sites assessed by the health care provider performing the dressing change using the Face, Legs, Activity, Cry, Consolability (FLACC) scale. The scale is scored in a range of 0-10 with 0 representing no pain.
Time Frame: Up to Week 4
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Blinding Effectiveness by Asking the Blinded Evaluator Which Treatment They Think the Donor Sites (A and B) Received
Description: Blinding effectiveness by asking the Blinded Evaluator which treatment they think the donor sites (A and B) received
Time Frame: Week 4 and 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 52 Weeks
Groups:
- Experimental: All Participants (Within Patient Control): Every subject received both interventions (RECELL and CONTROL) such that each subject served as their own control.
  RECELL + Telfa™ Clear and Xeroform™ dressings
  RECELL® Autologous Cell Harvesting Device: Application of RES prepared using the RECELL® Autologous Cell Harvesting Device along with Telfa™ Clear primary and Xeroform™ secondary wound dressings
  Telfa™ Clear and Xeroform™ dressings: Telfa™ Clear and Xeroform™ dressings
Arm/Group | Experimental: All Participants (Within Patient Control)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: All Participants (Within Patient Control) (N=3)
Graft Loss 135cm2 (Injury, poisoning and procedural complications) | 1 (1) — Graft loss due to shearing of a non-study site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03624192/Prot_SAP_001.pdf